CLINICAL TRIAL: NCT01404026
Title: Cortical Modulation With Transcranial Direct Current Stimulation (tDCS) for Neuropathic Symptoms Following Burn Injury.
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Neuropathic Symptoms Due to Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010-p-001209
Record Dates: First submitted 2011-06-29; First posted 2011-07-27 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pain; Burn Injury
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Pain; Burns | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Subjects will undergo 20 minutes of active tDCS stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Subjects will undergo sham tDCS stimulation, where the current is only active for 30 seconds.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Subjects will undergo tDCS stimulation. For both active and sham stimulation we will use electrodes at 35cm^2, with an intensity of 2mA. The anodal electrode will be placed over the primary motor cortex, and the cathode will be placed over the contralateral supraorbital area. For active stimulation, the current will be active for the duration of 20 minutes. For sham stimulation, the current will only be active for 30 seconds, simulating the sensations of active stimulation.
  Other Names: low intensity 1x1 direct current stimulator

SUMMARY:
The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) on the neuropathic symptoms (pain/itch) due to a burn injury. The investigators hypothesize that the active tDCS group will show a significant pain/itch reduction when compared to sham stimulation.

ELIGIBILITY:
STUDY ELIGIBILITY CRITERIA:

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. Any size closed wound from burn injury, occurring at least 3 weeks prior to enrollment in the study.

   - Subjects with burns in scalp area will be excluded from the study as the electrode may cause irritation to the injuries
4. Use of regular medications for pain and/or itching control at stable doses for at least 3 weeks prior to enrollment in the study
5. No contraindications to tDCS:

   * metallic implants in the head
   * implanted brain medical devices
6. Subject is not pregnant at the time of enrollment
7. Neuropathic pain or itching (rated at least 4 on the VAS) within the burn scar or donor site, (pain can be described as burning, stabbing, piercing, pins and needles, tearing sensation) for at least 3 weeks.

Please note: If a patient reports pain and itching, we will enroll the patient based upon their most dominant symptom.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effect of tDCS on pain/itch perception | Measured for approximately 2 weeks
  Determine whether active tDCS offers a greater benefit on pain reduction in patients with neuropathic symptoms (itch/pain) following burns as compared with sham tDCS. We hypothesize that active tDCS will be associated with a larger pain/itch reduction, as indexed by the Visual Analogue Scale for Pain/Itch (VAS). The subject's VAS score will be measured immediately before the tDCS stimulation sessions and after the tDCS stimulation sessions for the duration of their participation in the trial.

SECONDARY OUTCOMES:
Effect of tDCS on motor cortex excitability | Measured for approximately 2 weeks.
  To investigate whether active tDCS induces changes in motor cortex and spinal cord excitability as indexed by single and paired-pulse transcranial magnetic stimulation (TMS) as compared with sham tDCS. We will also determine whether these changes are correlated with the clinical outcome (pain/itch reduction). The subject's cortical excitability will be measured immediately before the tDCS stimulation sessions and after the tDCS stimulation sessions for the duration of their participation in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States